CLINICAL TRIAL: NCT04129021
Title: High Resolution and High Speed Multimodal Ophthalmic Imaging
Brief Title: High Resolution, High-speed Multimodal Ophthalmic Imaging
Acronym: IMA-MODE
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Centre Hospitalier National d'Ophtalmologie des Quinze-Vingts (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: P19-03; 2019-A00942-55 (Registry Identifier: N° IDRCB)
Record Dates: First submitted 2019-08-19; First posted 2019-10-16 (Actual); Last update posted 2025-11-18 (Actual); Status verified 2025-11

CONDITIONS: Retinitis Pigmentosa; Maculopathy, Age Related; Macular Dystrophy; Macular Edema; Retinal Detachment; Retinal Degeneration; Glaucoma; Vascular Inflammation; Hypertension; Stroke; Diabetes; Corneal Dystrophy; Keratoconus; Dry Eye; Trauma
MeSH Terms: conditions — Retinitis Pigmentosa; Macular Degeneration; Macular Edema; Retinal Detachment; Retinal Degeneration; Glaucoma; Hypertension; Stroke; Diabetes Mellitus; Corneal Dystrophies, Hereditary; Keratoconus; Dry Eye Syndromes; Wounds and Injuries

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- High-resolution retinal imaging through adaptive optics (Experimental): High-resolution retinal imaging through adaptive optics, full field OCT and holographic systems
  Interventions: Device: High-resolution retinal imaging through adaptive optics; Device: High-resolution retinal imaging through holographic systems

INTERVENTIONS:
Device: High-resolution retinal imaging through adaptive optics — The protocol consists of performing retinal imaging using full-field optical coherence tomography. The participant is asked to put his forehead against the temple supports and his chin on a chin rest. The subject will be asked to fix a test pattern in the form of a cross. The pattern is positioned according to the desired eccentricity with respect to the fovea. The actual acquisition lasts a few seconds, possibly repeated to cover the field of the desired eye. The acquisition protocol depends on the subjects, their pathology and the system used; the area examined will be modified on a case by case basis. The total duration of each exam can be estimated at less than half an hour, with frequent breaks.
Device: High-resolution retinal imaging through holographic systems — The protocol consists of performing retinal imaging using a laser Doppler holography. For each system, the participant is asked to put his forehead against the temple supports and his chin on a chin rest. The subject will be asked to fix a test pattern in the form of a cross. The pattern is positioned according to the desired eccentricity with respect to the fovea. The actual acquisition lasts a few seconds, possibly repeated to cover the field of the desired eye. The acquisition protocol depends on the subjects, their pathology and the system used; the area examined will be modified on a case by case basis. The total duration of each exam can be estimated at less than half an hour, with frequent breaks.

SUMMARY:
Knowledge of the pathogenesis of ocular conditions, a leading cause of blindness, has benefited greatly from recent advances in ophthalmic imaging. However, current clinical imaging systems are limited in resolution, speed, or access to certain structures of the eye.

The use of a high-resolution imaging system improves the resolution of ophthalmoscopes by several orders of magnitude, allowing the visualization of many microstructures of the eye: photoreceptors, vessels, nerve bundles in the retina, cells and nerves in the cornea.

The use of a high-speed acquisition imaging system makes it possible to detect functional measurements such as the speed of blood flow. The combination of data from multiple imaging systems to obtain multimodal information is of great importance for improving the understanding of structural changes in the eye during a disease.

The purpose of this project is to observe structures that are not detectable with routinely used systems.

DETAILED DESCRIPTION:
The goal of the project is the capture and analysis of images with the IMA-MODE systems, in order to evaluate the performance of these systems compared to the existing clinical imaging devices used at the National Hospital of Ophthalmology.

This project should identify the best techniques to image the eye, and select the most promising techniques to evolve towards a possible development of a medical device.

ELIGIBILITY:
Inclusion Criteria:

* People over 18
* Patient with a pathology affecting the eye or healthy volunteer
* Participant who signed the consent
* Beneficiaries of the health insurance

Exclusion Criteria:

* Patients with a history of photosensitivity.
* Patients who have just received a photodynamic therapy treatment (
* Patients taking drugs with photosensitivity as a side effect.
* Persons with pacemakers or other implanted electronic medical device
* Patients with viral conjunctivitis or any other infectious disease.
* Patients with skin lesions on the neck or forehead
* Patients at high risk of damage from optical radiation, such as aphakic patients, or patients with decreased sensitivity to light due to fundus disease.
* Pregnant or lactating women
* Participant unable to be followed throughout the study
* Vulnerable people
* Subjects with predisposition to closure of the iridocorneal angle

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 1200 (Estimated)
Dates: Start 2019-07-03 (Actual); Primary Completion 2027-07 (Estimated); Study Completion 2027-07 (Estimated)

PRIMARY OUTCOMES:
Visualization of a structure of interest and measuring the short-term and long-term reproducibility of the data collected compared to routine systems | From date of inclusion until the date of last documented progression , assessed up to 5 years
  Obtain the visualization of a structure of interest or obtain a measurement that are not detectable with the systems used routinely by analyzing images with image analysis software dedicated by a multidisciplinary group including doctors and physicists, assisted by computer scientists
  The visualization of the structure of interest in at least one area of the image will be considered the main criterion of success.

CONTACTS AND LOCATIONS:
Overall Officials: Michel PAQUES, Principal Investigator — Centre Hospitalier National d'Ophtalmologie des Quinze-Vints
Locations (1):
- Centre Hospitalier National d'Ophtalmologie des Quinze-Vingts, Paris, France

REFERENCES:
- [Derived] Paques M, Norberg N, Chaumette C, Sennlaub F, Rossi E, Borella Y, Grieve K. Long Term Time-Lapse Imaging of Geographic Atrophy: A Pilot Study. Front Med (Lausanne). 2022 Jun 22;9:868163. doi: 10.3389/fmed.2022.868163. eCollection 2022. PMID 35814763